CLINICAL TRIAL: NCT05076110
Title: Nonopioid Pain Control Regimen After Arthroscopic Hip Procedures
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kelechi R. Okoroha, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-003441
Record Dates: First submitted 2021-09-29; First posted 2021-10-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Hip Arthroscopy
MeSH Terms: interventions — Oxycodone; Ibuprofen; Gabapentin; Acetaminophen; Methocarbamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care Group (Active Comparator): Subjects will receive standard of care pain medication Oxycodone for pain control following hip arthroscopy procedure
  Interventions: Drug: Oxycodone
- Non-Opiate Pain Control Group (Experimental): Subjects will receive a non-opiate pain control regime using Ibuprofen, Gabapentin, Acetaminophen, Methocarbamol for pain control following hip arthroscopy procedure.
  Interventions: Drug: Ibuprofen; Drug: Gabapentin; Drug: Acetaminophen; Drug: Methocarbamol

INTERVENTIONS:
Drug: Oxycodone — 5 mg tablets every 4 hours postoperatively as needed for pain control
  Arms: Standard of Care Group
Drug: Ibuprofen — 800 mg three times a day for 2 weeks postoperatively for pain control; not to exceed 3200 mg/day
  Arms: Non-Opiate Pain Control Group
Drug: Gabapentin — 300 mg three times a day for 5 days then wean off by day 10 postoperatively
  Arms: Non-Opiate Pain Control Group
Drug: Acetaminophen — 1000 mg three times a day for up to 4 weeks postoperatively for pain control; not to exceed 4 grams per day
  Arms: Non-Opiate Pain Control Group
Drug: Methocarbamol — 500 mg three times a week for 2 weeks postoperatively
  Other Names: Robaxin
  Arms: Non-Opiate Pain Control Group

SUMMARY:
This study is being conducted to evaluate the effectiveness of post-operative pain control without using narcotic pain medications.

ELIGIBILITY:
Inclusion Criteria:

• Scheduled for a primary Hip Arthroscopy at Mayo Clinic (Rochester, MN)

Exclusion Criteria:

* medical history of known allergies or intolerance to allergies or intolerance to Motrin, Gabapentin, Tylenol, dexamethasone, tramadol, or Robaxin.
* Substantial alcohol or drug abuse.
* History of narcotics within 6 months of surgery.
* Pregnancy.
* Renal impairment.
* Peptic ulcer disease.
* GI bleeding.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 188 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in pain score | Baseline, 14 days post-operatively
  Measure using a visual analog scale (VAS) to rate pain on a scale 0-10; 0=no pain to 10=worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Kelechi Okoroha, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No